CLINICAL TRIAL: NCT00994747
Title: Sensitive Periods in Early Flavor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Julie A. Mennella, Member, Monell Chemical Senses Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 803712
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: infancy; nutrition; protein hydrolysate formula; flavor preferences; food preferences; growth; emotional development; mother-infant interaction; infant temperament; feeding patterning; taste receptor and obesity genotype; sensitive period
MeSH Terms: conditions — Food Preferences | interventions — pregestimil; Flavoring Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group EEEEEEE (Active Comparator): Infant is fed Enfamil from 0.5-7.5 months of life
  Interventions: Other: Enfamil, milk-based formula
- Group ENEEEEE (Experimental): Infant is fed Enfamil during 0.5-1.5 months of life, Nutramigen from 1.5-2.5 months of life and then Enfamil 2.5-7.5 of life.
  Interventions: Other: Nutramigen (Flavor and Type of Infant Formula)
- Group EENEEEE (Experimental): Infant is fed Enfamil 0.5-2.5 months of life, Nutramigen from 2.5-3.5 months of life and then Enfamil from 3.5 to 7.5 months of life
  Interventions: Other: Nutramigen (Flavor and Type of Infant Formula)
- Group EEENEEE (Experimental): Infant is fed Enfamil from 0.5-3.5 months of life, Nutramigen from 3.5-4.5 months of life and then Enfamil from 4.5-7.5 months of life.
  Interventions: Other: Nutramigen (Flavor and Type of Infant Formula)
- Group ENNNEEE (Experimental): Infant if fed Enfamil from month 0.5-1.5 months of life, Nutramigen from 1.5 to 3.5 months of life and then Enfamil again 3.5-7.5 months of life.
  Interventions: Other: Nutramigen (Flavor and Type of Infant Formula)
- Group NNNNNNN (Experimental): Infant is fed Nutramigen from 0.5-7.5 months of life.
  Interventions: Other: Nutramigen (Flavor and Type of Infant Formula)

INTERVENTIONS:
Other: Nutramigen (Flavor and Type of Infant Formula) — Nutramigen, protein hydrolysate formula, fed to infants as sole formula source during specified times during the first 8.5 months of life
  Arms: Group EEENEEE; Group EENEEEE; Group ENEEEEE; Group ENNNEEE; Group NNNNNNN
Other: Enfamil, milk-based formula — Enfamil, milk-based formula, fed as formula source during first 8.5 months of life
  Arms: Group EEEEEEE

SUMMARY:
Flavor is the primary dimension by which young children determine food acceptance. However, children are not merely miniature adults since sensory systems mature postnatally and their responses to certain tastes differ markedly from adults. Moreover, emerging research has revealed that there are sensitive periods during infancy such that early flavor experiences serve to modify later responses to flavors and foods. The proposed study aims to investigate this important issue by using as a model system a class of infant formulas which are hydrolyzed protein based and thus have very pronounced and distinctive flavors which are unpalatable to older-aged infants and adults. This research was initiated because of anecdotal reports by pediatricians that although it is easy to introduce this type of formula to infants during the first months of life, it becomes extremely difficult to do so later in infancy. Indeed, recent studies in the investigators' laboratory provided the first experimental demonstration that infants younger than 4 months of age willingly accept substantial amounts of, and satiate while feeding, a novel, protein hydrolysate formula. In marked contrast, infants older than 4 months reject the protein hydrolysate formula and this rejection occurs within the first minute of a feed, a finding that strongly suggests the sensory qualities of the formula are responsible, at least in part, for this rejection. Moreover, this rejection is not evident when the investigators test older-aged infants with other unfamiliar, but non-hydrolysate, formulas. In other words, the rejection appears to be in response to a particular component or components of protein hydrolysate formulas. This shift in acceptability can be ameliorated by prior exposure. That is, if these formulas are introduced to infants within the first few months of life and are fed continuously, they remain highly acceptable throughout infancy and early childhood. These observations implicate a sensitive period during development, occurring somewhere before 4 months of age, during which exposure to a formula, which is unpalatable to adults and infants over 4 months of age without exposure, renders it acceptable and presumably palatable. To the investigators' knowledge, this is the clearest example of a sensitive period in the development of responses to foods and flavors in humans thus far identified.

There is a paucity of information on whether and how the composition of formulas fed to infants influences their short-term feeding behaviors during the first few months of life. The primary objective of this longitudinal study is to determine the period during early infancy when exposure to the casein-hydrolysate formula, Nutramigen, renders it acceptable during later infancy. The study also aims to determine how early sensory experiences with formula impact upon food acceptance during infancy (8-9 months of age) and childhood. The investigators will also explore how variation in the genes that encode for taste receptors influence preferences for foods and other behaviors.

DETAILED DESCRIPTION:
This is a basic research, longitudinal and experimental study in which infants will be randomized into one of six groups (N=10-15 per group) differing in the timing and type of formula that the infant will be fed during each month of the 7-month exposure period. Each mother-infant dyad will be studied from the 2-3rd week of life until approximately 9 months of age. When the infant is less than three weeks of age and the mother's decision to formula feed is well established, infants will be randomized into one of six groups differing in the timing and type of formula that the infant will be fed during each month of the 7-month exposure period. One group (Control EEEEEEE) will be assigned to a milk-based formula, Enfamil (E), whereas another group (NNNNNNN) will be assigned to Nutramigen (N) during the entire 7-month period of this study. The other 4 groups will be assigned to feed Nutramigen for specified periods during their first seven months of life (Groups ENEEEEE, EEENEEE, ENNNEEE).

A variety of methodologies developed in our laboratory will be employed to capture the infants' responses to a particular flavor or taste after the exposure period. That is, at the end of the exposure period, infants will be videotaped while they are 1) feeding formulas; 2) feeding foods (e.g., cereal; soups) that differ in flavors; and 3) exploring scented toys. Each month, infants will be weighed and measured for length as well as evaluated for cognitive and motor development and mothers will completed standardized questionnaires regarding infant temperament. A cheek swab from the mothers and infants will be obtained and genotyped for taste receptor and taste- and obesity- related genes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infants of any racial background
* Infants may be of either sex
* Infants must be 2 weeks of age
* Infants must be exclusively feeding a cow's milk-based formula
* Mothers must be over 18 years of age

Exclusion Criteria:

* Infants who were preterm
* Infants who have medical conditions that interfere with feeding or eating
* No major complications during pregnancy or at birth

Ages: 2 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2006-11; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
infants' intake, length of feeding and patterning of feeding of Nutramigen relative to Enfamil (infant-led feeding condition) | 0.5-8.5 months

SECONDARY OUTCOMES:
infant growth (weight and length) | 0.5 to 8.5 months of life
maternal perceptions of infant enjoyment of feeding | 8.5 months
infants' exploration of toys as a function of scent | 9 months
infants' intake of foods as a function of flavor and chemical composition | 8 months and 2-3 years
infants' temperament and behavioral development | 0.5 months -2years
taste receptor and obesity genotypes. | 8 months and 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Mennella, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Mennella JA, Lukasewycz LD, Castor SM, Beauchamp GK. The timing and duration of a sensitive period in human flavor learning: a randomized trial. Am J Clin Nutr. 2011 May;93(5):1019-24. doi: 10.3945/ajcn.110.003541. Epub 2011 Feb 10. PMID 21310829
- [Result] Mennella JA, Ventura AK, Beauchamp GK. Differential growth patterns among healthy infants fed protein hydrolysate or cow-milk formulas. Pediatrics. 2011 Jan;127(1):110-8. doi: 10.1542/peds.2010-1675. Epub 2010 Dec 27. PMID 21187303
- [Derived] Mennella JA, Trabulsi JC, Papas MA. Effects of cow milk versus extensive protein hydrolysate formulas on infant cognitive development. Amino Acids. 2016 Mar;48(3):697-705. doi: 10.1007/s00726-015-2118-7. Epub 2015 Oct 26. PMID 26497857